CLINICAL TRIAL: NCT03751267
Title: Effects of Paediatric Tuina (Massage) on Constipation and Related Symptoms Among the Pre-school Aged Children - a Randomized Control Trial
Brief Title: Effects of Paediatric Tuina (Massage) on Constipation and Related Symptoms Among the Pre-school Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW18-132
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2018-11

CONDITIONS: Constipation
Keywords: Paediatric Massage, Constipation, Pre-school Children
MeSH Terms: conditions — Constipation | interventions — Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuina (massage) (Experimental): Tuina is massage based on Traditional Chinese Medicine (TCM) principles.
  Interventions: Procedure: Tuina (massage)
- Wait-list control (No Intervention): This group of patients will receive Tuina (massage) 4 weeks after baseline assessments.

INTERVENTIONS:
Procedure: Tuina (massage) — Tuina is massage based on Traditional Chinese Medicine (TCM) principles.
  Arms: Tuina (massage)

SUMMARY:
The research is a collaborative project by HKU and Yan Chai Hospital, funded by Social Welfare Development Fund of HKSAR. The study is designed as a prospective randomized control trial with the primary objective to investigate the efficacy of pediatric tuina (massage) on the functional constipation of pre-school aged children.

Our study is a pragmatic research comparing the pediatrictuina(massage)treatment with care as usual, with the objectives of investigating

1. if a non-invasive, easy to learn pediatrictuina (massage) protocol could improve the constipation and related symptoms experienced by the pre-school age children
2. if there is a positive impact on the caregiver-children relationship and the children's behaviour (a sub-group analysis) when the constipation symptoms improved.

The subjects of this study are pre-school age children (age 2-6) who are serviced by Yan Chai Hospital Social Service Department (YCHSS).The subjects will be openly recruited through the service units serving pre-school aged children under YCHSS. Rome IV criteria will be used to identify the children who suffer from constipation.

I. Trial Design This is a multicentre, pragmatic randomized control trial (PRCT) with a prospective design

Hypothesis 1:

Applying regular pediatrictuina (massage) (3 times a week, for 4 weeks ) on pre-school aged children with functional constipation will improve one or more of the following symptoms.

* Frequency of defecations
* Episode of incontinence
* Excessive stool retention
* Painful or hard bowel movements
* Presence of a large fecal mass in the rectum that may obstruct the toilet

Hypothesis 2:

The stress level of the caregiver of the study subjects improve as the constipation syndrome of the subjects improve.

Hypothesis 3:

The children with behavior problem who suffered from constipation will have less behavior issue when their functional constipation syndromes improved

Total 160 pre-school aged children with functional constipation and their caregiver will be openly recruited from the institutions/service units operated by the pediatric service unit of Yan Chai Hospital Social Service Department.The recruited children must suffer from functional constipation symptoms (based on Rome IV criteria). All accepted subjects will be in dyad. (i.e. 1 pre-school aged child and his designated caregiver, who commits bring the child to attend all treatment and assessment sessions, respond to all caregivers' assessment and fill in the daily logbook).

All applications will be screened by the social workers in the centres based on the inclusion and exclusion criteria. Qualified applicants will be invited for a health assessment conducted by registered TCM practitioner in the research team to confirm their suitability and invite them to sign the consent form. The consented dyad will be allocated randomly into treatment group and waitlist control group.

II. Intervention A 10 minutes structured pediatric massage protocol with specific applications technique will be performed on the children allocated to the treatment group three times a week for 4 consecutive weeks by trained TCM practitioners in the service units of YCHSS. The caregivers of the children need to participate in all assessment sessions and fill in the log book provided.

In the 1st 4 weeks, the children in the waitlist control group will not receive any pediatrictuina (massage). After the dyad completed the assessment sessions at baseline and week 4 ,(served as Treatment-as-Usual Control), children in the control group will receive the same 4 weeks of pediatric massage as the treatment group. The data collected before the treatment begins at week 4 will serve as the 2nd baseline for the waitlist control group.

The treatment protocol involve 8 steps.The massage area focuses on the abdomen and lower back of the recipients. All the movements/steps selected are well established and commonly used in the TCM practices. Any movement that demand professional training or involve potential risk is excluded from the protocol.

III. Measurement of efficacy Efficacy of the treatments will be measured in multi dimensions before and after the treatment for both groups. The main outcome measures are defecation frequency per week, fecal incontinence frequency per week, and overall treatment success after 4 weeks intervention, 8 weeks intervention and 12 weeks (4 weeks after intervention stopped) Secondary outcome measures included

* abdominal pain and painful defecation based on bowel diary,
* the children's subjective level of pain during bowel movement,
* score of child behavior questionnaire and
* score of caregiver impact and burden

ELIGIBILITY:
Inclusion Criteria:

* a. Pre-school age children: Age 2-6 b. Gender: male or female c. Suffered from functional constipation (base on Rome IV criteria) d. Currently receiving rehabilitation service in the pediatric service unit run by Yan Chai Hospital Social Service Department (e.g. Early Education and Training Centre (EETC), Special Child Care Centre (SCCC), On site Pre-school Rehabilitation Service team.) e. The caregiver of the child is committed to participate in the research activities, include:
* bringing the child to attend the treatment sessions and present during the treatment
* observing and recording the constipation related symptom of the child during the study period and respond on the outcome measurement tools.

(The caregiver is preferred to be a family member, but could also be a child-care provider who live with the study subject.) f. The legal guardian of the study subject, and the caregiver both sign the consent form.

Exclusion Criteria:

* Children in the following situation will be excluded from the study:

  1. who has contra-indication of massage
  2. who is currently receiving massage as a regular therapy
  3. who is known to suffer from any physical (anatomical) or physiological (hormonal or other body chemistry) cause that leads to constipation symptoms

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Defecation frequency per week | baseline, change from baseline at 4th week; change from baseline at 8th week
  Defecation frequency per week
Fecal incontinence frequency per week | baseline, change from baseline at 4th week; change from baseline at 8th week.
  Fecal incontinence frequency per week
Overall treatment success after 4 weeks of treatment | baseline, change from baseline at 4th week; change from baseline at 8th week
  Treatment success was defined as bowel movements ≥ 3 times per week and fecal incontinence ≤ once per 2 weeks.

SECONDARY OUTCOMES:
Frequency of abdominal pain and painful defecation | baseline, change from baseline at 4th week; change from baseline at 8th week.
  Abdominal pain and painful defecation based on the bowel diary
Pictorial scale of pain intensity | baseline, change from baseline at 4th week; change from baseline at 8th week.
  The children's subjective level of pain during bowel movement in pictorial scale in a range of 0-10.with 0 as no pain and 10 as extremely painful
Strengths and Difficulties Questionnaire (SDQ) | baseline, change from baseline at 4th week; change from baseline at 8th week.
  SDQ is a brief emotional and behavioural screening questionnaire for children and young people. The tool can capture the perspective of the parents
  The 25 items in the SDQ comprise 5 scales of 5 items each. Each item score 0-2. For each of the 5 scales the score can range from 0 to 10 if all items were completed. All subscale except prosocial score added up to total difficulties score
  1. Emotional symptoms subscale
  2. Conduct problems subscale
  3. Hyperactivity/inattention subscale
  4. Peer relationships problem subscale
  5. Prosocial behaviour subscale
  For parent completed SDQ Total difficulties score Normal 0-13 Borderline 14-16 Abnormal 17-40 Emotional problems score Normal 0-3 Borderline 4 Abnormal 5-10 Conduct problems score Normal 0-2 Borderline 3 Abnormal 4-10 Hyperactivity score Normal 0-5 Borderline 6 Abnormal 7-10 Peer problems score Normal 0-2 Borderline 3 Abnormal 4-10 Prosocial score Normal 6-10 Borderline 5 Abnormal 0-4
Care-giver's perceived stress level in visual analogue scale | baseline, change from baseline at 4th week; change from baseline at 8th week.
  Score of care-giver's perceived stress level based on visual analogue scale in a range of 0-10, with 0 as no stress and 10 as very stressful

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No